CLINICAL TRIAL: NCT02311660
Title: Study of the Safety and Efficacy of Neurostimulation of the Cholinergic Anti-Inflammatory Pathway Using a Vagal Nerve Stimulation Device in Patients With Active Refractory Crohn's Disease
Brief Title: Vagus Nerve Stimulation in Crohn's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: SetPoint Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPM-007
Record Dates: First submitted 2014-12-03; First posted 2014-12-08 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- vagus nerve stimulation (Experimental): Patients will have an implanted vagus nerve stimulation device.
  Interventions: Device: Vagus Nerve Stimulation Device

INTERVENTIONS:
Device: Vagus Nerve Stimulation Device — Cyberonics VNS System

SUMMARY:
This is an open label interventional study using an implantable vagus nerve stimulation device in patients with Crohn's disease who have active disease despite treatment with a tumor necrosis factor (TNF) antagonist drug.

DETAILED DESCRIPTION:
This will be an open-label, multicenter study of the safety, biological activity and clinical outcomes of an active implantable VNS device in patients with active refractory CD.

Patients will sign informed consent prior to screening and will undergo all screening and baseline assessment procedures including endoscopy and endoscopic biopsy prior to planned VNS implantation date. Those who meet all of the inclusion criteria and none of the exclusion criteria will be considered enrolled and will be implanted.

After a minimum of 14 days following the implantation, patients will have their first in-clinic visit (Week 0 Visit), during which they will begin self-delivered once-daily stimulation using the VNS device.

Patients will return for weekly visits between Weeks 1-4, at which time outcomes and safety assessments will be taken. At each visit between weeks 1 and 4, an attempt will be made to increase the output current to the maximum level tolerated. At the Week 4 Visit, another attempt to increase the output current will be made and the daily stimulation time will in addition be incremented by 60 seconds to 2 minutes total.

At the Week 6 Visit safety and outcomes assessments will be taken and another attempt to increase the output current will be made, and the daily stimulation time will in addition be incremented to 5 minutes total.

Patients will return at Week 8, at which time safety and outcomes assessments will be taken. If the patient has not achieved a clinical remission by CDAI, the frequency of stimulations will increase from once daily to 4 times daily.

At Week 12, the patient will return for safety and outcomes assessments. The final study visit will be at the Week 16 Visit, at which time patients will have final primary endpoint safety and outcomes assessments, including a follow-up endoscopy with endoscopic biopsy. If patients terminate the study prior to week 16, every effort will be made to perform all Week 16 Visit procedures during an Early Termination Visit.

Patients who complete the study will have the option to enroll in a long-term extension study. If they do not wish to participate in the extension study they can opt to either have their device permanently inactivated and left in place or have the device surgically explanted.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18-75 years, inclusive
* Written informed consent prior to any of the screening procedures
* Diagnosis of Crohn's disease for more than 4 months prior to Week -4 Visit, with small bowel and/or colonic involvement
* Current evidence of moderately-to-severely active disease defined by a Week -4 Visit Crohn's Disease Activity Index (CDAI) score of 220 to 450, inclusive
* Simple Endoscopic Score for Crohn's Disease evaluation at baseline showing presence of a minimal ulcer score of 2 or 3 in at least 1 segment
* Levels of fecal calprotectin greater than or equal to 200 microgram/gram feces at Week -4 Visit
* History of inadequate response and/or intolerance or adverse events leading to discontinuation of one or more TNF-alpha inhibitors (e.g., infliximab, adalimumab, or certolizumab pegol), or vedolizumab
* Female subjects of child-bearing potential are eligible if not pregnant, not planning to become pregnant during the course of the study, and committed to use of contraceptive methods with a failure rate of less than 1 percent per year

Exclusion Criteria:

* Celiac disease
* Diagnosis of ulcerative or indeterminate colitis
* Enterocutaneous, abdominal or pelvic fistulae with abscesses, or fistulae likely to require surgery during the course of the study period
* Bowel surgery, other than appendectomy, within 12 weeks prior to Week -4 Visit and/or has planned surgery or deemed likely to need surgery for Crohn's disease during the study period
* Extensive colonic resection, subtotal or total colectomy
* Presence of ileostomies, colostomies or rectal pouches
* Fixed symptomatic stenoses of small bowel or colon
* History of more than 3 small bowel resections or diagnosis of short bowel syndrome
* Use of prohibited medications inside the specified washout period (prior to Week -4 Visit), and throughout the study. Prohibited medications include the following:

  * TNF antagonists and vedolizumab may continue throughout the study, but treatments should have been given at a stable dose for at least 6 months prior to the screening date and should be maintained at this level throughout the study
  * Use of any natalizumab within 8 weeks
  * Use of glucocorticoids at doses greater than 10 mg prednisone orally QD, or an equivalent dose of other oral or parenteral glucocorticoids within 4 weeks
  * Use of cyclosporine, tacrolimus, sirolimus or mycophenolate mofetil within 4 weeks
  * Use of intravenous antibiotics for Crohn's disease within 4 weeks
  * Use of tube or enteral feeding, or elemental diet within 2 weeks
  * Rectal Treatment: Use of 5-aminosalicylates or corticosteroid enemas or suppositories within 2 weeks
  * Azathioprine, 6-mercaptopurine and methotrexate can be continued throughout the trial. These medications must have been used for >12 weeks, at stable dose for at least 3 weeks prior to the Week -4 Visit.
* Leukocytopheresis or granulocytopheresis within 2 weeks prior to Week -4 Visit
* Positive immunoassay for Clostridium difficile at Week -4 Visit
* Known HIV infection
* Known active in infection with Hepatitis B Virus or Hepatitis C Virus
* Current evidence of, or has been treated for a malignancy within the past five years (other than localized basal cell or squamous cell skin cancer, cervical dysplasia, or any cancer which has been fully staged as in situ and has been fully resected)
* History of evidence of adenomatous colonic polyps that have not been removed.
* Use of any investigational product within 30 days prior to Week -4 Visit for small molecules, or 8 weeks prior for monoclonal antibodies
* Significant psychiatric disease or substance abuse
* History of unilateral or bilateral vagotomy
* History of recurrent vaso-vagal syncope episodes
* Known obstructive sleep apnea
* Known history of cardiac rhythm disturbances, atrio-ventricular block of greater than first degree, or cardiac conduction pathway abnormalities other than isolated right bundle branch block or isolated left anterior fascicle block
* Significant pharyngeal dysfunction or swallowing difficulties
* Pre-existing clinically significant vocal cord damage or hoarseness
* Previously implanted electrically active medical devices (e.g., cardiac pacemakers, automatic implantable cardioverter-defibrillators)
* Asthma or chronic obstructive pulmonary disease not controlled by medications, or any other disease causing clinically significant dyspnea at time of screening
* A greater than or equal to 40 pack-year smoking history
* Active peptic ulcer disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Crohn's Disease Activity Index | Week 16

SECONDARY OUTCOMES:
Simple Endoscopic Score for Crohn's Disease (SES-CD) | Week 16
Inflammatory Bowel Disease Questionnaire (IBDQ) | Week 16
Heart Rate Variability (HRV) | Week 16
Changes in Whole Blood Lipopolysaccharide-Induced TNF Release Assay | Week 16
Serum Inflammation Mediators using Meso Scale Discovery Inflammation Multiplex Assay | Week 16
  Change in level of each mediator from baseline to Week 16
Adverse Events | Week 16
Device Deficiencies meeting the event definition from EN ISO 14155:2011 | Week 16
  Number of events occurring between first use of the device and Week 16 Visit

CONTACTS AND LOCATIONS:
Overall Officials: Geert D'Haens, M.D., Ph.D., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (4):
- Clinical Hospital Dubrava, Zagreb, Croatia
- Humanitas Research Hospital, Milan, Italy
- Academic Medical Center, Amsterdam, Netherlands
- Karolinska University Hospital, Solna, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No